CLINICAL TRIAL: NCT06468384
Title: Sympatholytic Effects of High Thoracic Erector Spinae Plane Block: A Prospective Observational Study on Changes in Optic Nerve Sheath Diameter
Brief Title: Sympatholytic Effects of High Thoracic Erector Spinae Plane Block: Changes in Optic Nerve Sheath Diameter
Status: Not yet recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, ismet çopur, principal investigator, Pamukkale University
Other Study IDs: PAU-ANEST-SI-IC-01
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Parapsychology; Dental Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Undergoing Thoracic Erector Spinae Plane Block: The study focuses on a cohort of adult patients who are receiving the thoracic erector spinae plane (ESP) block for pain management. These patients include individuals experiencing pain in the shoulder, arm, or neck, as well as those with complex regional pain syndrome. The patients are generally healthy adults, categorized under ASA I-II (American Society of Anesthesiologists Physical Status Classification System). The primary aim of the study is to observe changes in optic nerve sheath diameter (ONSD) following the ESP block and to investigate the potential impact on the stellate ganglion. Data will be collected through clinical examinations and ultrasound performed before and after the ESP block procedure. The study aims to enhance understanding of the ESP block's safety and potential autonomic effects.
  Interventions: Procedure: thoracic erector spinae plane (ESP) block

INTERVENTIONS:
Procedure: thoracic erector spinae plane (ESP) block — The thoracic erector spinae plane (ESP) block is a regional anesthesia technique used for pain management in complex regional pain syndrome. This procedure involves injecting 20 ml of 0.25% bupivacaine into the deep layers of the erector spinae muscles. The patient is positioned appropriately, and the injection site is identified using anatomical landmarks and ultrasound guidance, at the T2 level. A needle is then inserted perpendicularly until it contacts the transverse process, at which point the local anesthetic is administered. The primary objective is to provide significant pain relief.

SUMMARY:
The thoracic erector spinae plane (ESP) block is suggested to potentially affect the stellate ganglion, a key component of the sympathetic nervous system, thereby influencing autonomic functions. Changes in optic nerve sheath diameter (ONSD) are used as indicators of intracranial pressure changes. This study aims to investigate the effects of the ESP block on ONSD, providing insights into its impact on the stellate ganglion and enhancing the understanding of the ESP block's safety and efficacy.

DETAILED DESCRIPTION:
The thoracic erector spinae plane (ESP) block is a regional anesthesia technique. This technique involves the injection of local anesthetics into the deep layers of the erector spinae muscles, blocking both somatic and visceral pain pathways. Although various studies have been conducted on the effectiveness of this technique in different clinical situations over the years, further research is needed to understand the precise mechanisms behind its neuroanatomical effects.

The stellate ganglion, an important component of the sympathetic nervous system, plays a crucial role in the regulation of several autonomic functions. It has been suggested that the ESP block may affect the stellate ganglion through its injection at the upper thoracic levels. Changes in the optic nerve sheath diameter (ONSD) have been used as an important indicator of intracranial pressure changes. Any potential changes in ONSD following stellate ganglion blockade could help elucidate the effects of the ESP block, thus aiding in the understanding of its safety and potential benefits for analgesia.

The aim of this study is to investigate the changes in optic nerve sheath diameter in patients undergoing the thoracic ESP block, which could provide more information on the impact of the ESP block on the stellate ganglion. By doing so, we aim to gain further insights into the potential analgesic effects and safety of the ESP block.

ELIGIBILITY:
Inclusion Criteria:

* Adults with neck, shoulder, and arm pain
* Those with complex regional pain syndrome

The study will include 15 adult patients who are planned to receive T2-ESP block treatment.

* Age between 18-65 years
* Both genders
* ASA physical status I-II

Exclusion Criteria:

* Those who refuse procedures and tests
* Individuals with conditions that can increase intracranial pressure
* Those with severe heart failure
* Individuals with second or third-degree atrioventricular block
* Those with a history of unstable angina
* Individuals with COPD or chronic asthma
* Those who have experienced a myocardial infarction (MI) within the last 6 weeks
* Individuals with a heart rate below 50 beats per minute
* Those with systolic blood pressure below 90 mmHg
* Individuals with liver failure
* Those with kidney failure
* Individuals for whom a supraclavicular block is anatomically impossible
* Those with neurological or psychological conditions that complicate test evaluation
* Individuals allergic to any of the study medications
* Pregnant individuals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adults with neck, shoulder, and arm pain
  * Those with complex regional pain syndrome
  The study will include 15 adult patients who are planned to receive T2-ESP block treatment.
  * Age between 18-65 years
  * Both genders
  * ASA physical status I-II
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter (ONSD) | Before the block and 30 minutes after the block.
  To investigate the change in optic nerve sheath diameter (ONSD) following the thoracic erector spinae plane (ESP) block.

SECONDARY OUTCOMES:
Pain relief Visual Analog Scale (VAS) | Pain levels will be assessed using the VAS before the block, 30 minutes after the block, and 24 hours later to evaluate the effectiveness of the intervention.
  The Visual Analog Scale (VAS) is a tool for measuring pain intensity, using a line marked with "no pain" (0) at one end and "worst pain imaginable" (10) at the other. Patients mark a point on the line that reflects their pain level, and the distance from the "no pain" end to the mark is recorded as the VAS score. This straightforward, subjective measure provides a quantitative assessment of pain, useful for tracking changes over time, evaluating treatment effectiveness, and enhancing communication between patients and healthcare providers.
Monitoring of Perfusion Index (PI) | All perfusion index (PI) values will be measured at 3-minute intervals using 2 pulse oximeter sensors on both the blocked and contralateral unblocked upper extremities up to 30 minutes after local anesthetic injection.
  The perfusion index (PI) is a numerical value that reflects the pulsatile blood flow in peripheral tissues, measured non-invasively using a pulse oximeter. It indicates the strength of the blood flow at the sensor site, providing valuable information about peripheral perfusion.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chin KJ, El-Boghdadly K. Mechanisms of action of the erector spinae plane (ESP) block: a narrative review. Can J Anaesth. 2021 Mar;68(3):387-408. doi: 10.1007/s12630-020-01875-2. Epub 2021 Jan 6. PMID 33403545
- [Result] Shirodkar CG, Munta K, Rao SM, Mahesh MU. Correlation of measurement of optic nerve sheath diameter using ultrasound with magnetic resonance imaging. Indian J Crit Care Med. 2015 Aug;19(8):466-70. doi: 10.4103/0972-5229.162465. PMID 26321806
- [Result] Kim E, Lim JA, Choi CH, Lee SY, Kwak S, Kim J. Assessment of the changes in cardiac sympathetic nervous activity using the pupil size changes measured in seated patients whose stellate ganglion is blocked by interscalene brachial plexus block. Korean J Anesthesiol. 2023 Apr;76(2):116-127. doi: 10.4097/kja.22324. Epub 2022 Oct 24. PMID 36274253
- [Result] Maissan IM, Dirven PJ, Haitsma IK, Hoeks SE, Gommers D, Stolker RJ. Ultrasonographic measured optic nerve sheath diameter as an accurate and quick monitor for changes in intracranial pressure. J Neurosurg. 2015 Sep;123(3):743-7. doi: 10.3171/2014.10.JNS141197. Epub 2015 May 8. PMID 25955869
- [Result] Kim MS, Yoon KB, Yoon DM, Kim DH. Effect of cervical sympathetic block on optic nerve sheath diameter measured by ultrasonography. Ultrasound Med Biol. 2015 Jun;41(6):1599-604. doi: 10.1016/j.ultrasmedbio.2015.01.025. Epub 2015 Mar 5. PMID 25747936
- [Result] Dautzenberg KHW, Zegers MJ, Bleeker CP, Tan ECTH, Vissers KCP, van Geffen GJ, van der Wal SEI. Unpredictable Injectate Spread of the Erector Spinae Plane Block in Human Cadavers. Anesth Analg. 2019 Nov;129(5):e163-e166. doi: 10.1213/ANE.0000000000004187. PMID 31107261
- [Result] Forero M, Peng P, Chan P. Horner syndrome following high thoracic erector spinae plane block. Can J Anaesth. 2022 Mar;69(3):400-401. doi: 10.1007/s12630-021-02177-x. Epub 2021 Dec 13. No abstract available. PMID 34902105
- [Result] Elkoundi A, Eloukkal Z, Bensghir M, Belyamani L. Priapism following erector spinae plane block for the treatment of a complex regional pain syndrome. Am J Emerg Med. 2019 Apr;37(4):796.e3-796.e4. doi: 10.1016/j.ajem.2019.01.012. Epub 2019 Jan 11. PMID 30660341
- [Result] Hong JH, Park JH, Park KB, Lee JY. Sympatholytic Effect of the High Thoracic Erector Spinae Plane Block. Pain Physician. 2024 Jan;27(1):43-49. PMID 38285034